CLINICAL TRIAL: NCT04021498
Title: Simvastatin in the Prevention of Recurrent Pancreatitis, a Triple Blind, Randomized Controlled Trial
Brief Title: Simvastatin in the Prevention of Recurrent Pancreatitis
Acronym: SIMBA-16
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Enrique de-Madaria (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other); Generalitat Valenciana (Other)
Responsible Party: Sponsor-Investigator, Enrique de-Madaria, Principal Investigator, Hospital General Universitario de Alicante
Organization: Hospital General Universitario de Alicante (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SIMBA-16
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Pancreatitis Relapsing
Keywords: Pancreatitis; Acute pancreatitis; Chronic pancreatitis; Simvastatin; Recurrent
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatitis; Recurrence | interventions — Simvastatin; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): placebo
  1 year
  Interventions: Other: Placebo
- Simvastatin (Experimental): 40 mg
  1 year
  Interventions: Drug: Simvastatin 40mg

INTERVENTIONS:
Drug: Simvastatin 40mg — phase III, triple-blind randomised placebo-controlled trial comparing simvastatin 40 mg/day versus placebo (lactose). One hundred and fifty eight patients with recurrent AP (at least 2 episodes) will be included (79 per arm of treatment). Treatment and follow-up will last for 12 months.
  Other Names: Brand name: Simvastatin Normon, 40 mg
  Arms: Simvastatin
Other: Placebo — phase III, triple-blind randomised placebo-controlled trial comparing simvastatin 40 mg/day versus placebo (lactose). One hundred and fifty eight patients with recurrent AP (at least 2 episodes) will be included (79 per arm of treatment). Treatment and follow-up will last for 12 months.
  Other Names: lactose (brand name: lactosa monohidrato Fagrón)
  Arms: Placebo

SUMMARY:
Recurrent acute pancreatitis and recurrent relapses of inflammation in chronic pancreatitis are an important problem. In some cases, prevention of these acute flares of inflammation is not possible. Population-based studies and meta-analysis of randomized controlled trials suggest that statins may decrease the incidence of acute pancreatitis. SIMBA aims to investigate the effect of simvastatin on the incidence of new episodes of pancreatitis in recurrent acute pancreatitis and chronic pancreatitis. This is a non-profit, researcher-driven placebo-controlled multicenter (27 Spanish centers) randomized controlled trial

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is the 3rd cause of hospital admission due to gastrointestinal disease. Approximately 20% of the patients will relapse after a first episode of AP. The low frequency of relapse in biliary AP is due to the high effectiveness of cholecystectomy but a first episode of AP due to alcoholic or other etiologies is associated with relapse in one every four patients. Currently, besides counselling for alcohol and tobacco abstinence, there is no specific medical treatment that changes the natural history of recurrent AP. Recurrent AP is an intermediary stage in the pathogenesis of chronic pancreatitis (CP) and a subset of recurrent AP patients during their natural course transition to CP (one every three patients). Forty-five percent of patients with CP experience intermittent flares of pain. Simvastatin has been associated to a decrease in the incidence of AP in a population-based study (Wu et al, Gut. 2015) and in a meta-analysis of randomized controlled trials (Preiss et al, JAMA 2012).

The main aim of SIMBA (SIMvastatin in the prevention of recurrent pancreatitis, a triple Blind rAndomized controlled multicenter trial) is to compare the recurrence rate of pancreatitis in patients with established recurrent pancreatitis (acute pancreatitis and acute flares in chronic pancreatitis) consuming simvastatin versus placebo.

The secondary aims are 1) to compare in patients with recurrent AP at the end of follow-up period the progression to chronic pancreatitis on imaging (calcifications and/or dilated ductal system), as well as endocrine and exocrine pancreatic function; 2) to compare the severity of recurrent pancreatitis between both treatment arms.

Design: SIMBA is a triple-blind randomized placebo-controlled, parallel-group, superiority multicenter (27 Spanish centers) trial. This final protocol (version 4) was finished on June 20th 2018.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>=18) patients
2. At least 2 episodes of acute pancreatitis or acute flares of chronic pancreatitis
3. Written consent to participate in the study

Exclusion Criteria:

1. <2 episodes of pancreatitis in the last 12 months.
2. Statin consumption in the previous year.
3. Contraindications to the use of Statins
4. Cholelithiasis or choledocholitiasis diagnosed in the last episode of pancreatitis
5. Endoscopic sphyncterotomy and/or cholecystectomy and/or pancreatic surgery between last episode of AP and recruitment or patients who are expected to undergo one of this techniques in less than a year.
6. Serum triglycerides >500 mg/dL without previous specific treatment before the last episode of pancreatitis, or in patients expected to have a change in their specific hypertriglyceridemia treatment in less than 1 year
7. Primary hyperparathyroidism that has been operated between last episode of pancreatitis and recruitment or will be operated in less than 1 year
8. Iatrogenic Pancreatitis
9. Abstinence syndrome due to alcohol or drugs and/or delirium tremens in the last 6 months before recruitment
10. Previous (last year) failure to attend follow-up medical visits, social problems that may be associated to failure to take the medication or to perform an adequate follow-up
11. Pregnancy, breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Primary end point | 1 year
  Recurrence of pancreatitis during the follow-up period. Pancreatitis is defined as 2 or more of the following criteria: I) increased amylase and/or lipase in blood higher than 3 times the upper limit of normality, II) typical abdominal pain and III) signs of acute pancreatitis or acute flare of inflammation in chronic pancreatitis on imaging (CT scan or MRI).

SECONDARY OUTCOMES:
Secondary end point | 1 year
  New-onset diabetes at the end of follow-up, according to the American Diabetes Association criteria. Blood levels of glycosylated hemoglobin at the end of follow-up will also be compared to baseline (beginning of the study)
New-onset exocrine pancreatic insufficiency | 1 year
  New-onset exocrine pancreatic insufficiency defined by fecal elastase-1 <100 mcg/g. Fecal elastase-1 levels at the end of follow-up will also be compared to baseline
Chronic Pancreatitis on imaging | 1 year
  Chronic Pancreatitis on imaging at the end of follow-up, defined as calcifications and/or dilated pancreatic duct (≥4mm) on a CT scan
All-cause hospital admissions | 1 year
  Frequency of all-cause hospital admissions
Severity of pancreatitis | 1 year
  Severity of pancreatitis according to the revision of the Atlanta Classification (moderate-to-severe versus mild)
Adherence to treatment | 1 year
  Percentage of the planned treatment consumed by the patient
Adverse events | 1 year
  Frequency of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Enrique de-Madaria, MD PhD, Principal Investigator — Gastroenterology Department, Hospital General Universitario de Alicante, Spain
Locations (1):
- Alicante, Alicante, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guilabert L, Cardenas-Jaen K, Vaillo-Rocamora A, Ruiz-Rebollo ML, Bolado-Concejo F, Martinez-Moneo E, Rivera-Irigoin R, Martin-Mateos R, Garcia-Rayado G, Lopez-Serrano A, Marti-Marques E, Rodriguez-Oballe JA, Francisco-Gonzalez M, Jimenez-Moreno MA, Canamares-Orbis P, Concepcion-Martin M, Pascual-Moreno I, Del Val A, Lauret-Brana E, Sanchez-Marin C, Del Pozo-Garcia AJ, Ledro-Cano D, Zapater P, Nunez-Otero J, Bernal-Lujan L, Singh VK, Papachristou GI, Garg PK, Wu BU, Mehta RM, de-Madaria E. Simvastatin in the prevention of recurrent pancreatitis: a triple-blinded randomised clinical trial (the SIMBA trial). Gut. 2026 Jan 2:gutjnl-2025-337154. doi: 10.1136/gutjnl-2025-337154. Online ahead of print. PMID 41482454
- [Derived] Cardenas-Jaen K, Vaillo-Rocamora A, Gracia A, Garg PK, Zapater P, Papachristou GI, Singh VK, Wu BU, de-Madaria E. Simvastatin in the Prevention of Recurrent Pancreatitis: Design and Rationale of a Multicenter Triple-Blind Randomized Controlled Trial, the SIMBA Trial. Front Med (Lausanne). 2021 Feb 10;7:494. doi: 10.3389/fmed.2020.00494. eCollection 2020. PMID 33644082